CLINICAL TRIAL: NCT05667701
Title: Soy Isoflavones For Inner City Infants At Risk For Asthma (SIRA) Study
Acronym: SIRA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Rajesh Kumar (Other)
Collaborators: Northwestern University (Other); University of South Florida (Other); University of Colorado, Denver (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor-Investigator, Rajesh Kumar, Professor of Pediatrics, Ann & Robert H Lurie Children's Hospital of Chicago
Organization: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAUSE-LCH-001; U01AI160018-01 (NIH)
Record Dates: First submitted 2022-12-20; First posted 2022-12-29 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Wheezing; Asthma in Children
Keywords: wheezing; soy isoflavone; PAI-1
MeSH Terms: conditions — Respiratory Sounds | interventions — Soybean Proteins

STUDY DESIGN:
Intervention Model Description: genotype stratified, quadruple blinded randomized clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Neither participants nor the clinical center investigators will be informed of the treatment group assignment to maintain the mask. The randomization sequence will be generated by the study statistician and uploaded to the REDCap database, and randomization will be implemented through REDCap. Only the treatment distribution center (study pharmacist) and the independent unblinded study statistician will have access to the actual treatment assignments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Soy isoflavone (Experimental): Soy isoflavone powder dosed in puree or liquid twice daily
  Interventions: Drug: Soy isoflavone
- Placebo (Placebo Comparator): Matching placebo powder dosed in puree or liquid twice daily
  Interventions: Drug: matching placebo

INTERVENTIONS:
Drug: Soy isoflavone — Soy isoflavone supplement (Novasoy) that contains isoflavones (genistein, daidzein, glycetein) given at a dose of genistein aglycone equivalents to provide the genistein dosing of 22.6 mg/day for children aged 2-10 months, and 30.3 mg/day children aged 10-24 months
  Other Names: Novasoy
  Arms: Soy isoflavone
Drug: matching placebo — A matching placebo also administered twice daily.
  Other Names: placebo
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to compare soy isoflavones to placebo in children who at risk of asthma and have a genetic variation which results in them making more of a pro-inflammatory protein, plasminogen activator inhibitor-1. The main questions this trail seeks to answer is: will soy isoflavones decrease the proportion of infants with aT2 high endotype at the end of treatment, and secondarily decrease the number of wheezing episodes in these children when given in the first year of life. Participants will be asked to ingest soy isoflavone or placebo twice daily mixed into a liquid or puree vehicle for 7 months from randomization. There will be 3 mandatory in-person visits, and 6 virtual visits in the first year. There will also be 11 monthly questionnaires and 1 in person visit in the observation year. Participants will have 4 nasal swabs, 3 blood draws, and also provide 4 stool samples over the course of the study.

DETAILED DESCRIPTION:
The study is designed as a single site, randomized, quadruple-masked, placebo-controlled, parallel group clinical trial. We will enroll 65 high risk infants with the PAI-1 risk genotype, who are less than 12 months of age, and will be randomized to one of two treatment groups. The treatment groups will be either oral isoflavone supplement (at doses similar to that seen in soy formula) or a matching placebo .

Screening will occur throughout each year, with genotyping occurring at the first visit, and assumption of care of individuals with the risk genotype after randomization. There will be a study run in period up to 12 months at which time subjects will be randomized. The treatment period will run for 7 months for each participant, and will have a 1 year observation period after the end of treatment.

At randomization, the investigators will assume the care of the children for all wheezing illnesses. The subjects will have either virtual or in person visits for each of the next 6 visits, followed by an in-person visit at the end of treatment. The subjects will also come in for in-person visits at times of viral illnesses. At randomization, end of treatment, viral illness, and end of study the subjects will have nasal swabs and nasosorption carried out. Blood draws will occur at randomization, end of treatment, and the end of study visit. Stool will be collected for microbiome assessment at randomization, the 3rd or 4th month of treatment, the end of treatment, and the end of the study at the end of the observation year. The study will also measure infant pulmonary function using a wearable device to assess expiratory variability overnight. This will be measured at randomization, viral illness, end of treatment, and at the end of the study after the 1 year observation period. The treatment period will run for 7 months for each participant, with a 1 year observation period after this.

ELIGIBILITY:
Inclusion Criteria:

1. Parent/guardian must be an adult (≥18 years of age) and able to understand and provide informed consent.
2. Age: Term infants (≥37 weeks gestational age) less than 12 months of age at recruitment
3. High risk of asthma: As determined by one or more of the following:

   1. A history of uni- or bi-parental asthma with onset in childhood by parent self report, OR
   2. Uni- or bi-parental asthma with onset after childhood along with the presence of one or more other comorbid atopic condition including allergic rhinitis, atopic dermatitis, or food allergy, OR
   3. atopic dermatitis in the child determined by parent report of a physician diagnosis
4. Genotype: Either homozygous or heterozygous for the PAI-1 risk allele (i.e. 4G4G or 4G5G).
5. Have a primary place of residence in one of the pre-selected recruitment census tracts as outlined in the SIRA Manual of Operations (MOP).

   1. Participants who do not live in the pre-selected census tracts but live within the Office of Management and Budget (OMB) defined Metropolitan Statistical Area and have publicly funded health insurance will qualify for inclusion.

Exclusion Criteria:

1. 1. Inability or unwillingness of a parent or guardian to give written informed consent or comply with study protocol.
2. Parents who will not include either a puree or some form of bottle feeding such that the infant would be able to take the investigational product in a puree or a liquid (expressed breast milk, supplemental formula, or a small amount of water).
3. Currently on a soy based formula.
4. Breastfeeding mothers who are taking soy supplements or soy enriched foods more than 2 times a week and will not stop this level of ingestion while breastfeeding.
5. On treatment for recurrent wheezing such as regular inhaled steroids.
6. The infant may not have the following specific contraindications: known congenital thyroid disease, or a history of estrogen sensitive clinically relevant mutations in the family (such as BRCA1).
7. Medication use

   1. Maternal use of tamoxifen in pregnancy or if breastfeeding
   2. Use of immunomodulatory medications such at methotrexate, mycophenolate, azathioprine, or other immunomodulatory agent in the mother if breastfeeding or in the infant.
8. Use of another investigational agent in the last 30 days prior to randomization.
9. Current, parent reported, diagnosis of mental illness or current, diagnosed or self-reported drug or alcohol abuse (in the primary caregiver) that, in the opinion of the investigator, would interfere with the participant's ability to comply with study requirements.
10. Known allergy to soy protein (either by reported allergy or skin testing to soy prior to randomization) or reported allergy to NovaSoy, from which the investigational product is compounded.
11. The infant is currently participating in another asthma-related pharmaceutical study or intervention study or who have participated in another asthma-related pharmaceutical study or intervention study in the month prior to enrollment.
12. Past or current medical problems or findings from physical examination or laboratory testing that are not listed above, which, in the opinion of the investigator, may pose additional risks from participation in the study, may interfere with the participant's ability to comply with study requirements or that may impact the quality or interpretation of the data obtained from the study.
13. Infant requiring intubation prior to screening.
14. Infant requiring > 3 hospitalizations for asthma symptoms/ wheezing illness prior to screening.
15. Infant requiring > 3 five day bursts of oral steroid at least 14 days apart from each other prior to screening.
16. Any chronic condition requiring use of systemic corticosteroids or another immunomodulating agent at screening or before randomization, and during the course of the study.
17. Non-adherence:

    1. Inability / unwillingness of the parents to induce the infant to swallow study medication
    2. Unwillingness of the parents to allow the staff to perform baseline measurements
18. Living with a foster parent as a ward of the state.
19. Caregiver does not have access to a phone (needed for scheduling appointments or responding to questionnaires).
20. Plan(s) for the family to move from the area during the study period.
21. The infant's caretaker does not primarily speak English or Spanish.

In order to be eligible to continue in the study following screening visit A (V1) , an individual must meet all of the following additional randomization criteria:

1. Must be ≥4 months and <12 months of age at randomization
2. Must have either 4G/4G or 4G/5G genotype
3. Cannot have had a severe wheezing exacerbation requiring ICU admission between screening (V1) and randomization (V3)
4. Cannot have had more than two wheezing / "asthma" episodes (separated from each other by at least 14 days), each requiring at least a 5 day course of oral steroids in the time between screening visit A (V1) and randomization (V3).

Ages: 2 Months to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 65 (Estimated)
Dates: Start 2024-09-18 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
T2 endotype | From week 0 (randomization) to week 30 (end of treatment)
  This measure is determined by the proportion of subjects designated as having a T2 high endotype at the end of the treatment period (week 32) in the soy genistein vs placebo treatment arms.

SECONDARY OUTCOMES:
wheezing episodes | 7 months
  Number of episodes of wheezing - based on numbers of reported episodes of illness associated with wheezing over the treatment period.
Expiratory variability index | from week 0 (randomization) to week 30 (end of treatment) and from week 0 (randomization) to week 88 (end of study)
  Infant pulmonary function assessed by measurement of the Expiratory Variability Index change from baseline
safety and tolerability | from week 0 (randomization) to week 88 (end of study)
  Number and grade of adverse events by treatment arm

OTHER OUTCOMES:
Other measures of wheezing and respiratory morbidity | week 88 - end of study visit
  modified asthma predictive index at the end of the study
sensitization to allergens | Week 30 at the end of treatment
  The proportion of participants sensitized to indoor allergens (assessed by measurement of Dermatophygoides farinae, Dermatophygoides pteronyssinius, dog, cat, cockroach, mouse sIgE) and food allergens (milk, egg, peanut, wheat, and soy)
work disruption due to child's asthma | Week 0 to week 30
  The ratio of the work hours missed due to child's asthma over the numbers of work hours in the past 14 days in active vs placebo groups at each visit.
Daycare/ pre-school Absences due to the child's asthma | from randomization (week 0) to the end of treatment (week 30) and secondarily to the end of the observation period (week 88)
  The ratio of the number of school days missed over the number of school days in session in active vs placebo participants

CONTACTS AND LOCATIONS:
Overall Officials: Rajesh Kumar, MD, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (2):
- United States (2):
  - Ann and Robert H Lurie Childrens Hospital of Chicago, Chicago, Illinois
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: Yes
At present, the investigators plan to make deidentified data available as per NIH policy at 3 years after the completion of the study. This will not include any identifying information but will include all the primary outcome data and the participant individual level data that were included in the analyses including relevant covariates. It is planned that the investigators will use AccessClinicalData@NIAID for this purpose.
Supporting Information: Study Protocol
Time Frame: The investigators anticipate that data will be made publicly available 3 years after completion of the study.
Access Criteria: Investigators will be able to apply for use of the data and this will be reviewed by a committee, to prevent duplicative efforts.